CLINICAL TRIAL: NCT02448108
Title: Internet Psychotherapy for Treating Bipolar Disorder in Primary Care
Brief Title: Internet Psychotherapy for Bipolar Disorder in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Northwestern University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Holly Swartz, Professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 00085129000; R34MH107541 (NIH)
Record Dates: First submitted 2015-05-13; First posted 2015-05-19 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- i-IPSRT (Experimental): Participants randomized to this arm will complete bi-weekly i-IPSRT modules over the course of 12 weeks and they will track their mood and SRM's via smartphones or computer.
  Interventions: Behavioral: i-IPSRT
- i-IPSRT + CH (Experimental): Participants randomized to this arm will complete bi-weekly i-IPSRT modules over the course of 12 weeks and they will track their mood and SRM's via smartphones or computer. Additionally, i-IPSRT support will be delivered by Clinical Helpers, who will reach out to participants in this arm via 5-10 minute weekly phone calls.
  Interventions: Behavioral: i-IPSRT
- CC (Controlled Condition) (Other): Participants randomized to this arm will receive brief written psychoeducational material that includes information about social rhythm regularity. This information will be either mailed or e-mailed to them.
  Interventions: Other: Written Psychoeducation

INTERVENTIONS:
Behavioral: i-IPSRT — internet IPSRT (a form of psychotherapy for individuals with bipolar disorder) will be offered via 12 specially-designed modules.
  CH will have participated in a two day training about Bipolar Disorder and IPSRT.
  Other Names: i-IPSRT + CH
  Arms: i-IPSRT; i-IPSRT + CH
Other: Written Psychoeducation — Written material about the importance of social rhythm regularity to mood stability in bipolar disorder
  Arms: CC (Controlled Condition)

SUMMARY:
The investigators will conduct a small pilot study to test the feasibility and acceptability of treating bipolar disorder (BP) in primary care with online psychotherapy delivered both with and without telephone, text, and email support from a clinical helper (CH). The ultimate goal of this work is to provide preliminary data needed to design a larger scale effectiveness study of online psychotherapy for treating BP in primary care.

DETAILED DESCRIPTION:
Over a third of individuals with bipolar spectrum disorders (BP) are treated exclusively in primary care settings, and yet, primary care providers (PCPs) are ill-equipped to manage this complex and disabling illness. Medications, which can be prescribed by PCPs, hasten recovery from illness and improve long-term course of illness for those with BP, but relapse and residual symptoms are common when individuals are treated with pharmacotherapy alone. Best practices treatment for BP includes adjunctive, BP-specific psychotherapy as a key element of effective care. And yet, evidence-based BP-specific psychotherapies that engage and modify targets specific to BP are typically unavailable in primary care settings. Online interventions have the potential to overcome barriers to accessing evidence-based psychosocial treatments for BP in primary care. In other settings and with other populations, effectiveness of online interventions improved when human support/coaching (clinical helpers; CH) via text, email, and telephone was added to the intervention. Interpersonal and Social Rhythm Therapy (IPSRT) is a BP-specific psychotherapy that uses a problem-solving approach to help individuals regularize their social rhythms in order to entrain underlying disturbances in circadian and sleep/wake regulation, factors that are increasingly recognized as playing important roles in the pathogenesis of BP. Its primary behavioral target is regularity of daily routines such as sleep/wake cycle and mealtimes. This construct is measured by the validated Social Rhythm Metric (SRM). The current project seeks to develop and conduct initial testing of an online version of IPSRT (i-IPSRT) for use in primary care. We will (1) evaluate the feasibility and acceptability of supported and unsupported online psychotherapy interventions for BP in primary care (i-IPSRT and i-IPSRT plus CH) compared to Control Condition (CC), (2) examine whether i-IPSRT and i-IPSRT + CH engages its primary behavioral target as measured by the SRM, and (3) explore the impact of i-IPSRT, i-IPSRT + CH, and CC on symptoms and functioning over 12 weeks. Information from this study will inform a larger trial to test the effectiveness of these approaches in primary care. The public health impact of developing an effective, technology-enabled approach to delivering evidenced-based psychotherapy that targets specific, modifiable, behaviors for BP in primary care settings is substantial, offering the potential to reduce illness burden and improve outcomes for individuals with this disabling disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older;
* meet DSM 5 criteria for bipolar disorder I, II or Other Specified Bipolar and Related Disorder;
* using the SCID 5;
* score > or = to 9 on Patient Health Questionnaire-9 or score > or = 155 on Internal State Scale;
* receiving care from a Primary Care Physician in a designated study site;
* access to broadband Internet connection and telephone; and
* ability to read and speak English.

Exclusion Criteria:

* Self-reported visual impairment that would prevent completion of study procedures;
* Psychotic disorder, substance use disorder or current manic episode, which would deem participation in the study either inappropriate or dangerous;
* currently receiving specialty mental health services for bipolar disorder from a psychiatrist or therapist;
* planning to leave Primary Care Practice within next 3 months; and
* active suicidal ideation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Client-Satisfaction Questionnaire | Up to Week 12
  measure of client satisfaction
Social Rhythm Metric (measure of lifestyle regularity) | Up to 12 weeks
  measure of lifestyle regularity
Supportive Accountability Questionnaire | Up to Week 12
  assesses level of perceived accountability to another person for treatment participation

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptoms | up to 12 weeks
  measure of depressive symptoms
Internal State Scale | up to 12 weeks
  measure of mood symptoms
Short Form-12 | up to 12 weeks
  measure of overall health status
Functional Assessment Short Test | up to 12 weeks
  assessment of impairment in functioning

CONTACTS AND LOCATIONS:
Overall Officials: Holly A Swartz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States